CLINICAL TRIAL: NCT07254351
Title: Biomechanical Analysis of the Impact of Lower Limb Length Discrepancy on Hip and Lumbar Spine Joints in Children
Brief Title: Analysis of the Biomechanical Impact of Lower Limb Length Inequality in PEDiatrics
Acronym: ABILMI-PED
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0746; 2025-A01923-46 (Other: ID-RCB)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lower Limb Length Discrepancy (LLD) in Children
Keywords: EOS imaging; Biomechanics; Lower limb length discrepancy (LLD); Pediatric orthopedics; Force platform; limb length
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with lower limb length discrepancy (LLD): Pediatric patients aged 10-15 years with an anatomical LLD > 5 mm, evaluated in the routine pediatric orthopedic care pathway.
  Interventions: Radiation: EOS Imaging System; Device: Force Platform (Bertec®, integrated into EOS cabin)

INTERVENTIONS:
Radiation: EOS Imaging System — Low-dose biplanar radiographs of the whole body in standing position (EOS Imaging System). At baseline, two EOS acquisitions will be performed in static standing position : one without compensation (natural position) and one with temporary orthopedic compensation (shoe lift under the shorter limb). At 24 months, one EOS acquisition will be performed without compensation. Each acquisition lasts a few seconds, with radiation exposure 5 to 10 times lower than conventional radiographs.
Device: Force Platform (Bertec®, integrated into EOS cabin) — Ground reaction force (GRF) measurements obtained from a force platform integrated in the EOS cabin. The platform records weight distribution and center of pressure during static standing posture. Measurements are fully synchronized with EOS acquisitions, without additional time or discomfort for participants. At baseline, GRF measurements will be collected in two conditions (with and without orthopedic compensation). At 24 months, GRF measurements will be collected in the non-compensated condition.

SUMMARY:
Lower limb length discrepancy (LLD) is a frequent condition in pediatric orthopedics. Even moderate discrepancies can induce pelvic obliquity and compensatory scoliosis, modifying the distribution of joint loads at the hips and lumbar spine. These biomechanical imbalances are suspected to contribute to early degenerative conditions such as osteoarthritis or chronic low back pain.

The aim of this study is to quantify the biomechanical impact of LLD in children aged 10 to 15 years, using a combination of low dose biplanar EOS imaging (EOS Imaging System) and synchronized ground reaction force (GRF) measurements from integrated force platforms. These data will be used in musculoskeletal models developed in collaboration with the Biomechanics and Impact Mechanics Laboratory (LBMC, Laboratoire de Biomécanique et Mécanique des Chocs), enabling the estimation of hip joint and lumbar intervertebral disc loads.

This is the first pediatric study integrating EOS imaging, force platforms, and personalized musculoskeletal modeling to explore the mechanical consequences of LLD. The findings are expected to improve clinical reasoning and guide early therapeutic strategies.

DETAILED DESCRIPTION:
Lower limb length discrepancy (LLD) is a frequent condition in pediatric orthopedics. Even moderate discrepancies can induce pelvic obliquity and compensatory scoliosis, modifying the distribution of joint loads at the hips and lumbar spine. These biomechanical imbalances are suspected to contribute to early degenerative conditions such as osteoarthritis or chronic low back pain.

The aim of this study is to quantify the biomechanical impact of LLD in children aged 10 to 15 years, using a combination of low dose biplanar EOS imaging (EOS Imaging System) and synchronized ground reaction force (GRF) measurements from integrated force platforms. These data will be used in musculoskeletal models developed in collaboration with the Biomechanics and Impact Mechanics Laboratory (LBMC, Laboratoire de Biomécanique et Mécanique des Chocs), enabling the estimation of hip joint and lumbar intervertebral disc loads.

A temporary orthopedic compensation (shoe lift) will also be tested to assess its immediate biomechanical effect. Participants will be evaluated at baseline (two EOS acquisitions: with and without compensation) and at 2 years (without compensation).

This is the first pediatric study integrating EOS imaging, force platforms, and personalized musculoskeletal modeling to explore the mechanical consequences of LLD. The findings are expected to improve clinical reasoning and guide early therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10-15 years
* Anatomical LLD > 5 mm, clinically measured
* EOS imaging indicated by the pediatric orthopedic surgeon in routine care
* Ability to stand still for 30 seconds without assistance
* Covered by social security
* Parental consent and non-opposition obtained

Exclusion Criteria:

* - Functional or postural LLD without true anatomical discrepancy
* History of major pelvic or spinal surgery
* Severe neurological or orthopedic condition preventing standing (e.g. cerebral palsy, progressive myopathy)
* Fixed equinus deformity preventing plantar support
* Major lower limb deformity (severe genu varum/valgum)
* Contraindication or inability to undergo EOS imaging

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of approximately 100 pediatric patients (aged 10 to 15 years) presenting with an anatomical lower limb length discrepancy (LLD) greater than 5 mm, confirmed by clinical evaluation. Participants will be recruited consecutively during routine outpatient visits at the Pediatric Orthopedics Department of Hôpital Femme-Mère-Enfant (HFME), Hospices Civils de Lyon, Bron, France. This hospital is a tertiary referral center in pediatric orthopedics, receiving children from the Rhône-Alpes region and beyond.
  All included patients will undergo EOS imaging as part of their standard clinical assessment for LLD, ensuring that the study is fully integrated within the regular care pathway. The cohort therefore represents a specialized clinical sample of children with LLD, rather than a general population or community-based sample.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Asymmetry of Hip Joint Contact Forces (%) in Static Standing | At baseline (Day 0, without compensation)
  Hip joint contact force asymmetry index (%): calculated as AI (%) = 100 × (F_long - F_short) / [(F_long + F_short)/2], where F_long and F_short are side-specific resultant hip joint contact forces (estimated by musculoskeletal modeling from EOS imaging and ground reaction force data). Units: percent (%).Higher values indicate greater asymmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry HAUMONT, MD, Principal Investigator — Hospices Civils de Lyon

IPD SHARING:
Plan to Share IPD: No